CLINICAL TRIAL: NCT04216121
Title: Local AblativeTherapy for Oligoprogressive Non-Small-Cell Lung Cancer Treated With First-line OSImertinib
Brief Title: LAT for Oligoprogressive NSCLC Treated With First-line OSImertinib
Acronym: LAT-FLOSI
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S63270
Record Dates: First submitted 2019-12-09; First posted 2020-01-02 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Non-Small Cell Lung Cancer With Mutation in Epidermal Growth Factor Receptor
Keywords: First line osimertinib; Local ablative therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Local ablative therapy — Stereotactic body radiotherapy
  Other Names: SBRT
Procedure: Local ablative therapy — Surgery

SUMMARY:
To determine whether in patients with EGFR mutated advanced NSCLC and osimertinib as first-line treatment, the (repeated) use of LAT to ≤ 3 OP lesions and continuation of first-line osimertinib, improves the median progression-free survival by more than 3 months (i.e. PFS2-PFS1 = >3 months).

DETAILED DESCRIPTION:
The (repeated) use of LAT to ≤ 3 OP lesions with continuation of first-line osimertinib, is endorsed by international guidelines (NCCN, ESMO).

In this phase IIb prospective non-randomized observational trial, we want to document the benefit of LAT in this patient cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥ 18 years of age
2. Established histological diagnosis of advanced NSCLC, not suitable for radical treatment, with an EGFR actionable mutation receiving first-line targeted TKI therapy with osimertinib
3. Initial radiologically confirmed response (at least stable disease) to osimertinib assessed 3 months post commencing osimertinib according to RECIST criteria v1.1.
4. Confirmed OPD defined as ≤ 3 intra- and extracranial sites of progressive disease. OP may be defined as progression of an individual metastasis according to RECIST or on 2 consecutive imaging studies at least 2 months apart with a minimum of 5mm increase in size from baseline or an unambiguous development of a new metastatic lesion with a grand total of 3 lesions. All sites must be visible, imaging defined targets, not previously treated with radiation or radiofrequency and suitable for treatment with LAT as determined by the local multi-disciplinary team (MDT).
5. Adequate baseline organ function to allow LAT to all the OP targets.
6. Predicted life expectancy ≥ 6 months
7. Karnofsky Index ≥ 60% and ECOG 0-2
8. Provision of written informed consent
9. Female participants must be surgically sterile or postmenopausal if SBRT is planned to the abdominal area or must agree to use effective contraception during the period of therapy.

Exclusion Criteria:

1. > 3 sites of progressive disease
2. Oligoprogressive metastases not amenable to LAT
3. Radiotherapy or radiofrequency ablation near the OP lesion prior to the inclusion in the LAT-FLOSI study
4. Co-morbidities considered clinically precluding the safe use of LAT
5. Any psychological, sociological or geographical issue potentially hampering compliance with the study
6. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Established histological diagnosis of advanced NSCLC, not suitable for radical treatment, with an EGFR actionable mutation receiving first-line targeted TKI therapy with osimertinib. Confirmed oligoprogressive disease defined as ≤ 3 intra- and extracranial sites of progressive disease
Sampling Method: Probability Sample
Enrollment: 39 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
PFS 2 | Time from start of osimertinib until first PD after LAT or death whichever comes first, up to 3 year after LAT
  Progression Free Survival 2

SECONDARY OUTCOMES:
Time to next line systemic therapy | Time from LAT until initiation of next line systemic therapy or death whichever comes first, up to 3 years after LAT
Patterns of disease progression | Time from LAT until disease progression or death whichever comes first, up to 3 years after LAT
  Patterns of disease progression after local ablative therapy (LAT) identified on sequential CT scans taken at 3 monthly intervals to document the natual history of the disease after LAT
Radiotherapy induced toxicity | Change in toxicity measured from baseline up to 3 years after radiotherapy
  Acute and late radiotherapy induced toxicities assessed using the CTCAE v4.0. and the RTOG/EORTC late morbidity score. Acute events are defined as ≤ 90 days post SBRT and late events > 90 days.
Quality of life | Change in quality of life measured from baseline up to 3 years after radiotherapy
  Quality of life is measured by the EORTC QLQ-LC13 questionnaire comprised both of multi-item and single-item measures of lung cancer-associated symptoms (i.e. coughing, haemoptysis, dyspnoea and pain) and side-effects from conventional chemo- and radiotherapy (i.e. hair loss, neuropathy, sore mouth and dysphagia).

CONTACTS AND LOCATIONS:
Locations (1):
- UZLeuven, Leuven, Belgium